CLINICAL TRIAL: NCT02259621
Title: Neoadjuvant Nivolumab, or Nivolumab in Combination With Ipilimumab, in Resectable Non-Small-Cell Lung Cancer.
Brief Title: Neoadjuvant Nivolumab, or Nivolumab in Combination With Ipilimumab, in Resectable NSCLC
Acronym: NA_00092076
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: J1414; NA_00092076 (Other: JHMIRB)
Record Dates: First submitted 2014-09-18; First posted 2014-10-08 (Estimated); Results first posted 2024-03-20 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; Carboplatin; Paclitaxel; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm B- Nivolumab (Experimental): Nivolumab administration:
  Three doses of nivolumab will be administered to enrolled patients on Day -42, Day -28, and Day-14 (+/- two days) prior to planned surgery on Day 0 or up to +10 days.
  Interventions: Drug: Nivolumab
- Arm C- Nivolumab, Carboplatin, & Paclitaxel (Experimental): Nivolumab 360 mg IV, Carboplatin AUC 5 or 6 IV, and Paclitaxel 175 or 200 mg/m2 IV every 21 days for 3 cycles prior to planned surgery on Day 0.
  Interventions: Drug: Nivolumab; Drug: Carboplatin; Drug: Paclitaxel
- Arm A- Nivolumab and Ipilimumab (Experimental): One dose of Nivolumab 3mg/kg IV & Ipilimumab 1mg/kg will be administered to enrolled patients on Day-42, then 2 doses of Nivolumab 3mg/kg will be administered to enrolled patients on Day-28 and Day-14
  Interventions: Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Nivolumab — Anti-PD-1 Therapy
  Other Names: BMS-936558 or MDX1106
Drug: Carboplatin — Anti-PD-1 Therapy
  Other Names: Paraplatin
  Arms: Arm C- Nivolumab, Carboplatin, & Paclitaxel
Drug: Paclitaxel — Anti-PD-1 Therapy
  Other Names: Taxol; Onxal
  Arms: Arm C- Nivolumab, Carboplatin, & Paclitaxel
Drug: Ipilimumab — Anti-PD-1 Therapy
  Arms: Arm A- Nivolumab and Ipilimumab

SUMMARY:
The proposed study will evaluate the safety and feasibility of preoperative administration nivolumab +/- ipilimumab in patients with high-risk resectable NSCLC, and will facilitate a comprehensive exploratory characterization of the tumor immune milieu and circulating immune cells and soluble factors in these patients. Data obtained in this study will provide valuable information for planning further prospective clinical trials of anti-PD-1 and other immunotherapies in NSCLC, both in the peri-operative and advanced disease setting.

DETAILED DESCRIPTION:
The proposed study will evaluate the safety and feasibility of preoperative administration nivolumab +/- ipilimumab in patients with high-risk resectable NSCLC, and will facilitate a comprehensive exploratory characterization of the tumor immune milieu and circulating immune cells and soluble factors in these patients. Data obtained in this study will provide valuable information for planning further prospective clinical trials of anti-PD-1 and other immunotherapies in NSCLC, both in the peri-operative and advanced disease setting. Ultimately, it is highly desirable to discover prospective biomarkers of response and toxicity to allow patients with NSCLC who are most likely to derive benefit to receive anti-PD-1 treatment, and conversely to minimize the risk of toxicity and ineffective treatment for patients who are unlikely to benefit.

In addition, an amendment to this study allows evaluation of the combination of nivolumab and the anti-CTLA4 antibody, ipilimumab in the neoadjuvant setting for the treatment of resectable NSCLC. In a large, multicohort, phase 1 trial, the ORR to combination ipilimumab and nivolumab therapy in patients unselected by PD-L1 status ranged from 39-47%. Incidence of grade 3-4 toxicity ranged from 33-37% across the combination ipilimumab and nivolumab cohorts which compares favorably with the rates of toxicity due to platinum doublet chemotherapy in this disease setting.

The current amendment includes addition of a third arm (Arm C) combining nivolumab and platinum-doublet chemotherapy in the neoadjuvant setting.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven non-small-cell lung cancer (core biopsy required).

  * Squamous or non-squamous histology
  * Diagnostic core biopsy specimens must be reviewed by a faculty pathologist at SKCCC or MSKCC
  * Either a formalin fixed paraffin block or a minimum of fifteen 5-micron tissue sections (slides) of tumor biopsy sample must be available for biomarker evaluation (study pathologist must review for adequacy of sampling). This can be obtained from archived tissues, or from a new biopsy if needed.
* Stage - High risk NSCLC with resection option for potential cure, as assessed by a faculty surgeon at SKCCC or MSKCC. This may include clinical stage IB (≥4cm), II and IIIA(see Appendix A). Subjects with N3 nodal involvement are not included.

ECOG performance status 0-1

-Adequate organ function as follows:

* Leukocytes ≥ 2,000/mm3
* Absolute neutrophil count (ANC) ≥ 1000/mm3
* Platelet count ≥ 100,000/mm3
* Hemoglobin ≥ 9 g/dL
* Creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥40 mL/min (if using the Cockcroft-Gault formula below):

Female CrCl = (140 - age in years) x weight in kg x 0.85 72 x serum creatinine in mg/dL

Male CrCl = (140 - age in years) x weight in kg x 1.00 72 x serum creatinine in mg/dL

* Total Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
* AST(SGOT), ALT(SGPT), and alkaline phosphatase ≤ 3 times the upper limit of normal
* Subjects must have adequate lung function to permit surgical resection determined by pre-enrollment pulmonary function tests to include DLCO

  * The effects of nivolumab on the developing human fetus are unknown. For this reason, women of child-bearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and for up to 23 weeks after the last dose of nivolumab. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Sexually active fertile men must use effective barrier birth control if their partners are WOCBP for up to 31 weeks after the last dose of nivolumab. WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within two weeks of registration. Women must not be breastfeeding.
  * Patient understands the study regimen, its requirements, risks and discomforts and is able and willing to sign the informed consent form. Voluntary signed and dated IRB/IEC approved written informed consent form in accordance with regulatory and institutional guidelines must be obtained before the performance of any protocol related procedures that are not part of normal patient care. Subjects must be competent to report AEs, understand the drug dosing schedule and use of medications to control AEs.

Exclusion Criteria:

* Subjects are excluded if they have an active, known or suspected autoimmune disease. Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger.
* Subjects are excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. As there is potential for hepatic toxicity with nivolumab or nivolumab/ipilimumab combinations, drugs with a predisposition to hepatoxicity should be used with caution in patients treated with nivolumab-containing regimen.
* Administration of chemotherapy or any other cancer therapy in the pre-operative period.
* Subjects with active concurrent malignancies are excluded i.e. cancers other than NSCLC (except non melanoma skin cancers, in situ bladder, gastric, breast, colon or cervical cancers/dysplasia).
* Subjects with brain metastasis are excluded from this study, and all patients should have brain imaging (either MRI brain or CT brain with contrast) prior to enrollment.
* Subjects with a history of symptomatic interstitial lung disease.
* Active systemic infection requiring therapy, positive tests for Hepatitis B surface antigen or Hepatitis C ribonucleic acid (RNA).
* Known positive history or positive test for Human Immunodeficiency Virus or Acquired ImmunoDeficiency Syndrome (AIDS).
* History of allergy to study drug components.
* Women who are pregnant or nursing.
* Men with female partners (WOCBP) that are not willing to use contraception.
* Prior therapy with an anti-PD-1, anti-PD-L1, anti-PDL-2, or anti-CTLA-4 antibody (or any other antibody targeting T cell co-regulatory pathways).
* Underlying medical conditions that, in the Investigator's opinion, will make the administration of study drug hazardous or obscure the interpretation of toxicity or adverse events.
* Prisoners or subjects who are involuntarily incarcerated or compulsorily detained for treatment of either a psychiatric or physical (e.g. infectious disease) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-09; Primary Completion 2022-10-14 (Actual); Study Completion 2027-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Forde, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (5):
- United States (4):
  - Johns Hopkins at Bayview Medical Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Memorial Sloan Kettering, New York, New York
  - Swedish Cancer Insitute, Edmonds, Washington
- Johnathan Spicer, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang X, Schwartz JC, Guo X, Bhatia S, Cao E, Lorenz M, Cammer M, Chen L, Zhang ZY, Edidin MA, Nathenson SG, Almo SC. Structural and functional analysis of the costimulatory receptor programmed death-1. Immunity. 2004 Mar;20(3):337-47. doi: 10.1016/s1074-7613(04)00051-2. PMID 15030777
- [Background] Dong H, Strome SE, Salomao DR, Tamura H, Hirano F, Flies DB, Roche PC, Lu J, Zhu G, Tamada K, Lennon VA, Celis E, Chen L. Tumor-associated B7-H1 promotes T-cell apoptosis: a potential mechanism of immune evasion. Nat Med. 2002 Aug;8(8):793-800. doi: 10.1038/nm730. Epub 2002 Jun 24. PMID 12091876
- [Background] Thompson RH, Kuntz SM, Leibovich BC, Dong H, Lohse CM, Webster WS, Sengupta S, Frank I, Parker AS, Zincke H, Blute ML, Sebo TJ, Cheville JC, Kwon ED. Tumor B7-H1 is associated with poor prognosis in renal cell carcinoma patients with long-term follow-up. Cancer Res. 2006 Apr 1;66(7):3381-5. doi: 10.1158/0008-5472.CAN-05-4303. PMID 16585157
- [Background] Topalian SL, Hodi FS, Brahmer JR, Gettinger SN, Smith DC, McDermott DF, Powderly JD, Carvajal RD, Sosman JA, Atkins MB, Leming PD, Spigel DR, Antonia SJ, Horn L, Drake CG, Pardoll DM, Chen L, Sharfman WH, Anders RA, Taube JM, McMiller TL, Xu H, Korman AJ, Jure-Kunkel M, Agrawal S, McDonald D, Kollia GD, Gupta A, Wigginton JM, Sznol M. Safety, activity, and immune correlates of anti-PD-1 antibody in cancer. N Engl J Med. 2012 Jun 28;366(26):2443-54. doi: 10.1056/NEJMoa1200690. Epub 2012 Jun 2. PMID 22658127
- [Background] Brahmer J, Reckamp KL, Baas P, Crino L, Eberhardt WE, Poddubskaya E, Antonia S, Pluzanski A, Vokes EE, Holgado E, Waterhouse D, Ready N, Gainor J, Aren Frontera O, Havel L, Steins M, Garassino MC, Aerts JG, Domine M, Paz-Ares L, Reck M, Baudelet C, Harbison CT, Lestini B, Spigel DR. Nivolumab versus Docetaxel in Advanced Squamous-Cell Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Jul 9;373(2):123-35. doi: 10.1056/NEJMoa1504627. Epub 2015 May 31. PMID 26028407
- [Background] Borghaei H, Paz-Ares L, Horn L, Spigel DR, Steins M, Ready NE, Chow LQ, Vokes EE, Felip E, Holgado E, Barlesi F, Kohlhaufl M, Arrieta O, Burgio MA, Fayette J, Lena H, Poddubskaya E, Gerber DE, Gettinger SN, Rudin CM, Rizvi N, Crino L, Blumenschein GR Jr, Antonia SJ, Dorange C, Harbison CT, Graf Finckenstein F, Brahmer JR. Nivolumab versus Docetaxel in Advanced Nonsquamous Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Oct 22;373(17):1627-39. doi: 10.1056/NEJMoa1507643. Epub 2015 Sep 27. PMID 26412456
- [Background] Gettinger S, Rizvi NA, Chow LQ, Borghaei H, Brahmer J, Ready N, Gerber DE, Shepherd FA, Antonia S, Goldman JW, Juergens RA, Laurie SA, Nathan FE, Shen Y, Harbison CT, Hellmann MD. Nivolumab Monotherapy for First-Line Treatment of Advanced Non-Small-Cell Lung Cancer. J Clin Oncol. 2016 Sep 1;34(25):2980-7. doi: 10.1200/JCO.2016.66.9929. Epub 2016 Jun 27. PMID 27354485
- [Background] Chen L. Co-inhibitory molecules of the B7-CD28 family in the control of T-cell immunity. Nat Rev Immunol. 2004 May;4(5):336-47. doi: 10.1038/nri1349. No abstract available. PMID 15122199
- [Background] Dunn GP, Bruce AT, Ikeda H, Old LJ, Schreiber RD. Cancer immunoediting: from immunosurveillance to tumor escape. Nat Immunol. 2002 Nov;3(11):991-8. doi: 10.1038/ni1102-991. PMID 12407406
- [Background] Retsas S, Priestman TJ, Newton KA, Westbury G. Evaluation of human lymphoblastoid interferon in advanced malignant melanoma. Cancer. 1983 Jan 15;51(2):273-6. doi: 10.1002/1097-0142(19830115)51:23.0.co;2-k. PMID 6821816
- [Background] West WH, Tauer KW, Yannelli JR, Marshall GD, Orr DW, Thurman GB, Oldham RK. Constant-infusion recombinant interleukin-2 in adoptive immunotherapy of advanced cancer. N Engl J Med. 1987 Apr 9;316(15):898-905. doi: 10.1056/NEJM198704093161502. PMID 3493433
- [Background] Tao MH, Levy R. Idiotype/granulocyte-macrophage colony-stimulating factor fusion protein as a vaccine for B-cell lymphoma. Nature. 1993 Apr 22;362(6422):755-8. doi: 10.1038/362755a0. PMID 8469286
- [Background] Phan GQ, Attia P, Steinberg SM, White DE, Rosenberg SA. Factors associated with response to high-dose interleukin-2 in patients with metastatic melanoma. J Clin Oncol. 2001 Aug 1;19(15):3477-82. doi: 10.1200/JCO.2001.19.15.3477. PMID 11481353
- [Background] Joseph RW, Sullivan RJ, Harrell R, Stemke-Hale K, Panka D, Manoukian G, Percy A, Bassett RL, Ng CS, Radvanyi L, Hwu P, Atkins MB, Davies MA. Correlation of NRAS mutations with clinical response to high-dose IL-2 in patients with advanced melanoma. J Immunother. 2012 Jan;35(1):66-72. doi: 10.1097/CJI.0b013e3182372636. PMID 22130161
- [Background] Kantoff PW, Higano CS, Shore ND, Berger ER, Small EJ, Penson DF, Redfern CH, Ferrari AC, Dreicer R, Sims RB, Xu Y, Frohlich MW, Schellhammer PF; IMPACT Study Investigators. Sipuleucel-T immunotherapy for castration-resistant prostate cancer. N Engl J Med. 2010 Jul 29;363(5):411-22. doi: 10.1056/NEJMoa1001294. PMID 20818862
- [Background] Hodi FS, O'Day SJ, McDermott DF, Weber RW, Sosman JA, Haanen JB, Gonzalez R, Robert C, Schadendorf D, Hassel JC, Akerley W, van den Eertwegh AJ, Lutzky J, Lorigan P, Vaubel JM, Linette GP, Hogg D, Ottensmeier CH, Lebbe C, Peschel C, Quirt I, Clark JI, Wolchok JD, Weber JS, Tian J, Yellin MJ, Nichol GM, Hoos A, Urba WJ. Improved survival with ipilimumab in patients with metastatic melanoma. N Engl J Med. 2010 Aug 19;363(8):711-23. doi: 10.1056/NEJMoa1003466. Epub 2010 Jun 5. PMID 20525992
- [Background] Krummel MF, Allison JP. CD28 and CTLA-4 have opposing effects on the response of T cells to stimulation. J Exp Med. 1995 Aug 1;182(2):459-65. doi: 10.1084/jem.182.2.459. PMID 7543139
- [Background] Leach DR, Krummel MF, Allison JP. Enhancement of antitumor immunity by CTLA-4 blockade. Science. 1996 Mar 22;271(5256):1734-6. doi: 10.1126/science.271.5256.1734. PMID 8596936
- [Background] Nishimura H, Honjo T. PD-1: an inhibitory immunoreceptor involved in peripheral tolerance. Trends Immunol. 2001 May;22(5):265-8. doi: 10.1016/s1471-4906(01)01888-9. PMID 11323285
- [Background] Freeman GJ, Long AJ, Iwai Y, Bourque K, Chernova T, Nishimura H, Fitz LJ, Malenkovich N, Okazaki T, Byrne MC, Horton HF, Fouser L, Carter L, Ling V, Bowman MR, Carreno BM, Collins M, Wood CR, Honjo T. Engagement of the PD-1 immunoinhibitory receptor by a novel B7 family member leads to negative regulation of lymphocyte activation. J Exp Med. 2000 Oct 2;192(7):1027-34. doi: 10.1084/jem.192.7.1027. PMID 11015443
- [Background] Latchman Y, Wood CR, Chernova T, Chaudhary D, Borde M, Chernova I, Iwai Y, Long AJ, Brown JA, Nunes R, Greenfield EA, Bourque K, Boussiotis VA, Carter LL, Carreno BM, Malenkovich N, Nishimura H, Okazaki T, Honjo T, Sharpe AH, Freeman GJ. PD-L2 is a second ligand for PD-1 and inhibits T cell activation. Nat Immunol. 2001 Mar;2(3):261-8. doi: 10.1038/85330. PMID 11224527
- [Background] Carter L, Fouser LA, Jussif J, Fitz L, Deng B, Wood CR, Collins M, Honjo T, Freeman GJ, Carreno BM. PD-1:PD-L inhibitory pathway affects both CD4(+) and CD8(+) T cells and is overcome by IL-2. Eur J Immunol. 2002 Mar;32(3):634-43. doi: 10.1002/1521-4141(200203)32:33.0.CO;2-9. PMID 11857337
- [Background] Chemnitz JM, Parry RV, Nichols KE, June CH, Riley JL. SHP-1 and SHP-2 associate with immunoreceptor tyrosine-based switch motif of programmed death 1 upon primary human T cell stimulation, but only receptor ligation prevents T cell activation. J Immunol. 2004 Jul 15;173(2):945-54. doi: 10.4049/jimmunol.173.2.945. PMID 15240681
- [Background] Sheppard KA, Fitz LJ, Lee JM, Benander C, George JA, Wooters J, Qiu Y, Jussif JM, Carter LL, Wood CR, Chaudhary D. PD-1 inhibits T-cell receptor induced phosphorylation of the ZAP70/CD3zeta signalosome and downstream signaling to PKCtheta. FEBS Lett. 2004 Sep 10;574(1-3):37-41. doi: 10.1016/j.febslet.2004.07.083. PMID 15358536
- [Background] Nishimura H, Nose M, Hiai H, Minato N, Honjo T. Development of lupus-like autoimmune diseases by disruption of the PD-1 gene encoding an ITIM motif-carrying immunoreceptor. Immunity. 1999 Aug;11(2):141-51. doi: 10.1016/s1074-7613(00)80089-8. PMID 10485649
- [Background] Nishimura H, Okazaki T, Tanaka Y, Nakatani K, Hara M, Matsumori A, Sasayama S, Mizoguchi A, Hiai H, Minato N, Honjo T. Autoimmune dilated cardiomyopathy in PD-1 receptor-deficient mice. Science. 2001 Jan 12;291(5502):319-22. doi: 10.1126/science.291.5502.319. PMID 11209085
- [Background] Wang J, Yoshida T, Nakaki F, Hiai H, Okazaki T, Honjo T. Establishment of NOD-Pdcd1-/- mice as an efficient animal model of type I diabetes. Proc Natl Acad Sci U S A. 2005 Aug 16;102(33):11823-8. doi: 10.1073/pnas.0505497102. Epub 2005 Aug 8. PMID 16087865
- [Background] Okazaki T, Tanaka Y, Nishio R, Mitsuiye T, Mizoguchi A, Wang J, Ishida M, Hiai H, Matsumori A, Minato N, Honjo T. Autoantibodies against cardiac troponin I are responsible for dilated cardiomyopathy in PD-1-deficient mice. Nat Med. 2003 Dec;9(12):1477-83. doi: 10.1038/nm955. Epub 2003 Nov 2. PMID 14595408
- [Background] Salama AD, Chitnis T, Imitola J, Ansari MJ, Akiba H, Tushima F, Azuma M, Yagita H, Sayegh MH, Khoury SJ. Critical role of the programmed death-1 (PD-1) pathway in regulation of experimental autoimmune encephalomyelitis. J Exp Med. 2003 Jul 7;198(1):71-8. doi: 10.1084/jem.20022119. PMID 12847138
- [Background] Blazar BR, Carreno BM, Panoskaltsis-Mortari A, Carter L, Iwai Y, Yagita H, Nishimura H, Taylor PA. Blockade of programmed death-1 engagement accelerates graft-versus-host disease lethality by an IFN-gamma-dependent mechanism. J Immunol. 2003 Aug 1;171(3):1272-7. doi: 10.4049/jimmunol.171.3.1272. PMID 12874215
- [Background] Konishi J, Yamazaki K, Azuma M, Kinoshita I, Dosaka-Akita H, Nishimura M. B7-H1 expression on non-small cell lung cancer cells and its relationship with tumor-infiltrating lymphocytes and their PD-1 expression. Clin Cancer Res. 2004 Aug 1;10(15):5094-100. doi: 10.1158/1078-0432.CCR-04-0428. PMID 15297412
- [Background] Thompson RH, Gillett MD, Cheville JC, Lohse CM, Dong H, Webster WS, Krejci KG, Lobo JR, Sengupta S, Chen L, Zincke H, Blute ML, Strome SE, Leibovich BC, Kwon ED. Costimulatory B7-H1 in renal cell carcinoma patients: Indicator of tumor aggressiveness and potential therapeutic target. Proc Natl Acad Sci U S A. 2004 Dec 7;101(49):17174-9. doi: 10.1073/pnas.0406351101. Epub 2004 Nov 29. PMID 15569934
- [Background] Ohigashi Y, Sho M, Yamada Y, Tsurui Y, Hamada K, Ikeda N, Mizuno T, Yoriki R, Kashizuka H, Yane K, Tsushima F, Otsuki N, Yagita H, Azuma M, Nakajima Y. Clinical significance of programmed death-1 ligand-1 and programmed death-1 ligand-2 expression in human esophageal cancer. Clin Cancer Res. 2005 Apr 15;11(8):2947-53. doi: 10.1158/1078-0432.CCR-04-1469. PMID 15837746
- [Background] Tsushima F, Tanaka K, Otsuki N, Youngnak P, Iwai H, Omura K, Azuma M. Predominant expression of B7-H1 and its immunoregulatory roles in oral squamous cell carcinoma. Oral Oncol. 2006 Mar;42(3):268-74. doi: 10.1016/j.oraloncology.2005.07.013. Epub 2005 Nov 3. PMID 16271509
- [Background] Thompson RH, Webster WS, Cheville JC, Lohse CM, Dong H, Leibovich BC, Kuntz SM, Sengupta S, Kwon ED, Blute ML. B7-H1 glycoprotein blockade: a novel strategy to enhance immunotherapy in patients with renal cell carcinoma. Urology. 2005 Nov;66(5 Suppl):10-4. doi: 10.1016/j.urology.2005.06.010. PMID 16194701
- [Background] Thompson RH, Gillett MD, Cheville JC, Lohse CM, Dong H, Webster WS, Chen L, Zincke H, Blute ML, Leibovich BC, Kwon ED. Costimulatory molecule B7-H1 in primary and metastatic clear cell renal cell carcinoma. Cancer. 2005 Nov 15;104(10):2084-91. doi: 10.1002/cncr.21470. PMID 16208700
- [Background] Dong H, Chen L. B7-H1 pathway and its role in the evasion of tumor immunity. J Mol Med (Berl). 2003 May;81(5):281-7. doi: 10.1007/s00109-003-0430-2. Epub 2003 Apr 30. PMID 12721664
- [Background] Azuma T, Yao S, Zhu G, Flies AS, Flies SJ, Chen L. B7-H1 is a ubiquitous antiapoptotic receptor on cancer cells. Blood. 2008 Apr 1;111(7):3635-43. doi: 10.1182/blood-2007-11-123141. Epub 2008 Jan 25. PMID 18223165
- [Background] Iwai Y, Terawaki S, Honjo T. PD-1 blockade inhibits hematogenous spread of poorly immunogenic tumor cells by enhanced recruitment of effector T cells. Int Immunol. 2005 Feb;17(2):133-44. doi: 10.1093/intimm/dxh194. Epub 2004 Dec 20. PMID 15611321
- [Background] Iwai Y, Ishida M, Tanaka Y, Okazaki T, Honjo T, Minato N. Involvement of PD-L1 on tumor cells in the escape from host immune system and tumor immunotherapy by PD-L1 blockade. Proc Natl Acad Sci U S A. 2002 Sep 17;99(19):12293-7. doi: 10.1073/pnas.192461099. Epub 2002 Sep 6. PMID 12218188
- [Background] Strome SE, Dong H, Tamura H, Voss SG, Flies DB, Tamada K, Salomao D, Cheville J, Hirano F, Lin W, Kasperbauer JL, Ballman KV, Chen L. B7-H1 blockade augments adoptive T-cell immunotherapy for squamous cell carcinoma. Cancer Res. 2003 Oct 1;63(19):6501-5. PMID 14559843
- [Background] Hirano F, Kaneko K, Tamura H, Dong H, Wang S, Ichikawa M, Rietz C, Flies DB, Lau JS, Zhu G, Tamada K, Chen L. Blockade of B7-H1 and PD-1 by monoclonal antibodies potentiates cancer therapeutic immunity. Cancer Res. 2005 Feb 1;65(3):1089-96. PMID 15705911
- [Background] Blank C, Brown I, Peterson AC, Spiotto M, Iwai Y, Honjo T, Gajewski TF. PD-L1/B7H-1 inhibits the effector phase of tumor rejection by T cell receptor (TCR) transgenic CD8+ T cells. Cancer Res. 2004 Feb 1;64(3):1140-5. doi: 10.1158/0008-5472.can-03-3259. PMID 14871849
- [Background] Scagliotti GV, Fossati R, Torri V, Crino L, Giaccone G, Silvano G, Martelli M, Clerici M, Cognetti F, Tonato M; Adjuvant Lung Project Italy/European Organisation for Research Treatment of Cancer-Lung Cancer Cooperative Group Investigators. Randomized study of adjuvant chemotherapy for completely resected stage I, II, or IIIA non-small-cell Lung cancer. J Natl Cancer Inst. 2003 Oct 1;95(19):1453-61. doi: 10.1093/jnci/djg059. PMID 14519751
- [Background] Arriagada R, Bergman B, Dunant A, Le Chevalier T, Pignon JP, Vansteenkiste J; International Adjuvant Lung Cancer Trial Collaborative Group. Cisplatin-based adjuvant chemotherapy in patients with completely resected non-small-cell lung cancer. N Engl J Med. 2004 Jan 22;350(4):351-60. doi: 10.1056/NEJMoa031644. PMID 14736927
- [Background] Douillard JY, Rosell R, De Lena M, Carpagnano F, Ramlau R, Gonzales-Larriba JL, Grodzki T, Pereira JR, Le Groumellec A, Lorusso V, Clary C, Torres AJ, Dahabreh J, Souquet PJ, Astudillo J, Fournel P, Artal-Cortes A, Jassem J, Koubkova L, His P, Riggi M, Hurteloup P. Adjuvant vinorelbine plus cisplatin versus observation in patients with completely resected stage IB-IIIA non-small-cell lung cancer (Adjuvant Navelbine International Trialist Association [ANITA]): a randomised controlled trial. Lancet Oncol. 2006 Sep;7(9):719-27. doi: 10.1016/S1470-2045(06)70804-X. PMID 16945766
- [Background] Waller D, Peake MD, Stephens RJ, Gower NH, Milroy R, Parmar MK, Rudd RM, Spiro SG. Chemotherapy for patients with non-small cell lung cancer: the surgical setting of the Big Lung Trial. Eur J Cardiothorac Surg. 2004 Jul;26(1):173-82. doi: 10.1016/j.ejcts.2004.03.041. PMID 15200998
- [Background] Butts CA, Ding K, Seymour L, Twumasi-Ankrah P, Graham B, Gandara D, Johnson DH, Kesler KA, Green M, Vincent M, Cormier Y, Goss G, Findlay B, Johnston M, Tsao MS, Shepherd FA. Randomized phase III trial of vinorelbine plus cisplatin compared with observation in completely resected stage IB and II non-small-cell lung cancer: updated survival analysis of JBR-10. J Clin Oncol. 2010 Jan 1;28(1):29-34. doi: 10.1200/JCO.2009.24.0333. Epub 2009 Nov 23. PMID 19933915
- [Background] Strauss GM, Herndon JE 2nd, Maddaus MA, Johnstone DW, Johnson EA, Harpole DH, Gillenwater HH, Watson DM, Sugarbaker DJ, Schilsky RL, Vokes EE, Green MR. Adjuvant paclitaxel plus carboplatin compared with observation in stage IB non-small-cell lung cancer: CALGB 9633 with the Cancer and Leukemia Group B, Radiation Therapy Oncology Group, and North Central Cancer Treatment Group Study Groups. J Clin Oncol. 2008 Nov 1;26(31):5043-51. doi: 10.1200/JCO.2008.16.4855. Epub 2008 Sep 22. PMID 18809614
- [Background] Pignon JP, Tribodet H, Scagliotti GV, Douillard JY, Shepherd FA, Stephens RJ, Dunant A, Torri V, Rosell R, Seymour L, Spiro SG, Rolland E, Fossati R, Aubert D, Ding K, Waller D, Le Chevalier T; LACE Collaborative Group. Lung adjuvant cisplatin evaluation: a pooled analysis by the LACE Collaborative Group. J Clin Oncol. 2008 Jul 20;26(21):3552-9. doi: 10.1200/JCO.2007.13.9030. Epub 2008 May 27. PMID 18506026
- [Background] NSCLC Meta-analyses Collaborative Group; Arriagada R, Auperin A, Burdett S, Higgins JP, Johnson DH, Le Chevalier T, Le Pechoux C, Parmar MK, Pignon JP, Souhami RL, Stephens RJ, Stewart LA, Tierney JF, Tribodet H, van Meerbeeck J. Adjuvant chemotherapy, with or without postoperative radiotherapy, in operable non-small-cell lung cancer: two meta-analyses of individual patient data. Lancet. 2010 Apr 10;375(9722):1267-77. doi: 10.1016/S0140-6736(10)60059-1. Epub 2010 Mar 24. PMID 20338627
- [Background] Burdett S, Stewart LA, Rydzewska L. A systematic review and meta-analysis of the literature: chemotherapy and surgery versus surgery alone in non-small cell lung cancer. J Thorac Oncol. 2006 Sep;1(7):611-21. PMID 17409927
- [Background] Depierre A, Milleron B, Moro-Sibilot D, Chevret S, Quoix E, Lebeau B, Braun D, Breton JL, Lemarie E, Gouva S, Paillot N, Brechot JM, Janicot H, Lebas FX, Terrioux P, Clavier J, Foucher P, Monchatre M, Coetmeur D, Level MC, Leclerc P, Blanchon F, Rodier JM, Thiberville L, Villeneuve A, Westeel V, Chastang C; French Thoracic Cooperative Group. Preoperative chemotherapy followed by surgery compared with primary surgery in resectable stage I (except T1N0), II, and IIIa non-small-cell lung cancer. J Clin Oncol. 2002 Jan 1;20(1):247-53. doi: 10.1200/JCO.2002.20.1.247. PMID 11773176
- [Background] Gilligan D, Nicolson M, Smith I, Groen H, Dalesio O, Goldstraw P, Hatton M, Hopwood P, Manegold C, Schramel F, Smit H, van Meerbeeck J, Nankivell M, Parmar M, Pugh C, Stephens R. Preoperative chemotherapy in patients with resectable non-small cell lung cancer: results of the MRC LU22/NVALT 2/EORTC 08012 multicentre randomised trial and update of systematic review. Lancet. 2007 Jun 9;369(9577):1929-37. doi: 10.1016/S0140-6736(07)60714-4. PMID 17544497
- [Background] Scagliotti GV, Pastorino U, Vansteenkiste JF, Spaggiari L, Facciolo F, Orlowski TM, Maiorino L, Hetzel M, Leschinger M, Visseren-Grul C, Torri V. Randomized phase III study of surgery alone or surgery plus preoperative cisplatin and gemcitabine in stages IB to IIIA non-small-cell lung cancer. J Clin Oncol. 2012 Jan 10;30(2):172-8. doi: 10.1200/JCO.2010.33.7089. Epub 2011 Nov 28. PMID 22124104
- [Background] Zitvogel L, Tesniere A, Kroemer G. Cancer despite immunosurveillance: immunoselection and immunosubversion. Nat Rev Immunol. 2006 Oct;6(10):715-27. doi: 10.1038/nri1936. Epub 2006 Sep 15. PMID 16977338
- [Background] Street SE, Cretney E, Smyth MJ. Perforin and interferon-gamma activities independently control tumor initiation, growth, and metastasis. Blood. 2001 Jan 1;97(1):192-7. doi: 10.1182/blood.v97.1.192. PMID 11133760
- [Background] Shankaran V, Ikeda H, Bruce AT, White JM, Swanson PE, Old LJ, Schreiber RD. IFNgamma and lymphocytes prevent primary tumour development and shape tumour immunogenicity. Nature. 2001 Apr 26;410(6832):1107-11. doi: 10.1038/35074122. PMID 11323675
- [Background] Al-Shibli KI, Donnem T, Al-Saad S, Persson M, Bremnes RM, Busund LT. Prognostic effect of epithelial and stromal lymphocyte infiltration in non-small cell lung cancer. Clin Cancer Res. 2008 Aug 15;14(16):5220-7. doi: 10.1158/1078-0432.CCR-08-0133. PMID 18698040
- [Background] Tormanen-Napankangas U, Soini Y, Paakko P. High number of tumour-infiltrating lymphocytes is associated with apoptosis in non-small cell lung carcinoma. APMIS. 2001 Jul-Aug;109(7-8):525-32. PMID 11552950
- [Background] Bremnes RM, Al-Shibli K, Donnem T, Sirera R, Al-Saad S, Andersen S, Stenvold H, Camps C, Busund LT. The role of tumor-infiltrating immune cells and chronic inflammation at the tumor site on cancer development, progression, and prognosis: emphasis on non-small cell lung cancer. J Thorac Oncol. 2011 Apr;6(4):824-33. doi: 10.1097/JTO.0b013e3182037b76. PMID 21173711
- [Background] Schneider T, Kimpfler S, Warth A, Schnabel PA, Dienemann H, Schadendorf D, Hoffmann H, Umansky V. Foxp3(+) regulatory T cells and natural killer cells distinctly infiltrate primary tumors and draining lymph nodes in pulmonary adenocarcinoma. J Thorac Oncol. 2011 Mar;6(3):432-8. doi: 10.1097/JTO.0b013e31820b80ca. PMID 21258248
- [Background] Shimizu K, Nakata M, Hirami Y, Yukawa T, Maeda A, Tanemoto K. Tumor-infiltrating Foxp3+ regulatory T cells are correlated with cyclooxygenase-2 expression and are associated with recurrence in resected non-small cell lung cancer. J Thorac Oncol. 2010 May;5(5):585-90. doi: 10.1097/JTO.0b013e3181d60fd7. PMID 20234320
- [Background] Woo EY, Yeh H, Chu CS, Schlienger K, Carroll RG, Riley JL, Kaiser LR, June CH. Cutting edge: Regulatory T cells from lung cancer patients directly inhibit autologous T cell proliferation. J Immunol. 2002 May 1;168(9):4272-6. doi: 10.4049/jimmunol.168.9.4272. PMID 11970966
- [Background] Zhang Y, Huang S, Gong D, Qin Y, Shen Q. Programmed death-1 upregulation is correlated with dysfunction of tumor-infiltrating CD8+ T lymphocytes in human non-small cell lung cancer. Cell Mol Immunol. 2010 Sep;7(5):389-95. doi: 10.1038/cmi.2010.28. Epub 2010 May 31. PMID 20514052
- [Background] Wong RM, Scotland RR, Lau RL, Wang C, Korman AJ, Kast WM, Weber JS. Programmed death-1 blockade enhances expansion and functional capacity of human melanoma antigen-specific CTLs. Int Immunol. 2007 Oct;19(10):1223-34. doi: 10.1093/intimm/dxm091. PMID 17898045
- [Background] Lynch TJ, Bondarenko I, Luft A, Serwatowski P, Barlesi F, Chacko R, Sebastian M, Neal J, Lu H, Cuillerot JM, Reck M. Ipilimumab in combination with paclitaxel and carboplatin as first-line treatment in stage IIIB/IV non-small-cell lung cancer: results from a randomized, double-blind, multicenter phase II study. J Clin Oncol. 2012 Jun 10;30(17):2046-54. doi: 10.1200/JCO.2011.38.4032. Epub 2012 Apr 30. PMID 22547592
- [Background] Wolchok JD, Hoos A, O'Day S, Weber JS, Hamid O, Lebbe C, Maio M, Binder M, Bohnsack O, Nichol G, Humphrey R, Hodi FS. Guidelines for the evaluation of immune therapy activity in solid tumors: immune-related response criteria. Clin Cancer Res. 2009 Dec 1;15(23):7412-20. doi: 10.1158/1078-0432.CCR-09-1624. Epub 2009 Nov 24. PMID 19934295
- [Background] Eggermont AM, Chiarion-Sileni V, Grob JJ, Dummer R, Wolchok JD, Schmidt H, Hamid O, Robert C, Ascierto PA, Richards JM, Lebbe C, Ferraresi V, Smylie M, Weber JS, Maio M, Konto C, Hoos A, de Pril V, Gurunath RK, de Schaetzen G, Suciu S, Testori A. Adjuvant ipilimumab versus placebo after complete resection of high-risk stage III melanoma (EORTC 18071): a randomised, double-blind, phase 3 trial. Lancet Oncol. 2015 May;16(5):522-30. doi: 10.1016/S1470-2045(15)70122-1. Epub 2015 Mar 31. PMID 25840693
- [Background] Carthon BC, Wolchok JD, Yuan J, Kamat A, Ng Tang DS, Sun J, Ku G, Troncoso P, Logothetis CJ, Allison JP, Sharma P. Preoperative CTLA-4 blockade: tolerability and immune monitoring in the setting of a presurgical clinical trial. Clin Cancer Res. 2010 May 15;16(10):2861-71. doi: 10.1158/1078-0432.CCR-10-0569. Epub 2010 May 11. PMID 20460488
- [Background] Woo SR, Turnis ME, Goldberg MV, Bankoti J, Selby M, Nirschl CJ, Bettini ML, Gravano DM, Vogel P, Liu CL, Tangsombatvisit S, Grosso JF, Netto G, Smeltzer MP, Chaux A, Utz PJ, Workman CJ, Pardoll DM, Korman AJ, Drake CG, Vignali DA. Immune inhibitory molecules LAG-3 and PD-1 synergistically regulate T-cell function to promote tumoral immune escape. Cancer Res. 2012 Feb 15;72(4):917-27. doi: 10.1158/0008-5472.CAN-11-1620. Epub 2011 Dec 20. PMID 22186141
- [Background] Chen H, Liakou CI, Kamat A, Pettaway C, Ward JF, Tang DN, Sun J, Jungbluth AA, Troncoso P, Logothetis C, Sharma P. Anti-CTLA-4 therapy results in higher CD4+ICOShi T cell frequency and IFN-gamma levels in both nonmalignant and malignant prostate tissues. Proc Natl Acad Sci U S A. 2009 Feb 24;106(8):2729-34. doi: 10.1073/pnas.0813175106. Epub 2009 Feb 6. PMID 19202079
- [Background] Liakou CI, Kamat A, Tang DN, Chen H, Sun J, Troncoso P, Logothetis C, Sharma P. CTLA-4 blockade increases IFNgamma-producing CD4+ICOShi cells to shift the ratio of effector to regulatory T cells in cancer patients. Proc Natl Acad Sci U S A. 2008 Sep 30;105(39):14987-92. doi: 10.1073/pnas.0806075105. Epub 2008 Sep 25. PMID 18818309
- [Background] Fu T, He Q, Sharma P. The ICOS/ICOSL pathway is required for optimal antitumor responses mediated by anti-CTLA-4 therapy. Cancer Res. 2011 Aug 15;71(16):5445-54. doi: 10.1158/0008-5472.CAN-11-1138. Epub 2011 Jun 27. PMID 21708958
- [Background] Taube JM, Anders RA, Young GD, Xu H, Sharma R, McMiller TL, Chen S, Klein AP, Pardoll DM, Topalian SL, Chen L. Colocalization of inflammatory response with B7-h1 expression in human melanocytic lesions supports an adaptive resistance mechanism of immune escape. Sci Transl Med. 2012 Mar 28;4(127):127ra37. doi: 10.1126/scitranslmed.3003689. PMID 22461641
- [Background] Schoenfeld J, Jinushi M, Nakazaki Y, Wiener D, Park J, Soiffer R, Neuberg D, Mihm M, Hodi FS, Dranoff G. Active immunotherapy induces antibody responses that target tumor angiogenesis. Cancer Res. 2010 Dec 15;70(24):10150-60. doi: 10.1158/0008-5472.CAN-10-1852. PMID 21159637
- [Derived] Zhang J, Ji Z, Caushi JX, El Asmar M, Anagnostou V, Cottrell TR, Chan HY, Suri P, Guo H, Merghoub T, Chaft JE, Reuss JE, Tam AJ, Blosser RL, Abu-Akeel M, Sidhom JW, Zhao N, Ha JS, Jones DR, Marrone KA, Naidoo J, Gabrielson E, Taube JM, Velculescu VE, Brahmer JR, Housseau F, Hellmann MD, Forde PM, Pardoll DM, Ji H, Smith KN. Compartmental Analysis of T-cell Clonal Dynamics as a Function of Pathologic Response to Neoadjuvant PD-1 Blockade in Resectable Non-Small Cell Lung Cancer. Clin Cancer Res. 2020 Mar 15;26(6):1327-1337. doi: 10.1158/1078-0432.CCR-19-2931. Epub 2019 Nov 21. PMID 31754049
- [Derived] Jafarnejad M, Gong C, Gabrielson E, Bartelink IH, Vicini P, Wang B, Narwal R, Roskos L, Popel AS. A Computational Model of Neoadjuvant PD-1 Inhibition in Non-Small Cell Lung Cancer. AAPS J. 2019 Jun 24;21(5):79. doi: 10.1208/s12248-019-0350-x. PMID 31236847
- [Derived] Cottrell TR, Thompson ED, Forde PM, Stein JE, Duffield AS, Anagnostou V, Rekhtman N, Anders RA, Cuda JD, Illei PB, Gabrielson E, Askin FB, Niknafs N, Smith KN, Velez MJ, Sauter JL, Isbell JM, Jones DR, Battafarano RJ, Yang SC, Danilova L, Wolchok JD, Topalian SL, Velculescu VE, Pardoll DM, Brahmer JR, Hellmann MD, Chaft JE, Cimino-Mathews A, Taube JM. Pathologic features of response to neoadjuvant anti-PD-1 in resected non-small-cell lung carcinoma: a proposal for quantitative immune-related pathologic response criteria (irPRC). Ann Oncol. 2018 Aug 1;29(8):1853-1860. doi: 10.1093/annonc/mdy218. PMID 29982279
- [Derived] Forde PM, Chaft JE, Smith KN, Anagnostou V, Cottrell TR, Hellmann MD, Zahurak M, Yang SC, Jones DR, Broderick S, Battafarano RJ, Velez MJ, Rekhtman N, Olah Z, Naidoo J, Marrone KA, Verde F, Guo H, Zhang J, Caushi JX, Chan HY, Sidhom JW, Scharpf RB, White J, Gabrielson E, Wang H, Rosner GL, Rusch V, Wolchok JD, Merghoub T, Taube JM, Velculescu VE, Topalian SL, Brahmer JR, Pardoll DM. Neoadjuvant PD-1 Blockade in Resectable Lung Cancer. N Engl J Med. 2018 May 24;378(21):1976-1986. doi: 10.1056/NEJMoa1716078. Epub 2018 Apr 16. PMID 29658848
- See also: Ferlay J, Shin HR, Bray F, Forman D, Mathers CD, Parkin D. GLOBOCAN 2008, Cancer Incidence and Mortality Worldwide: IARC CancerBase No. 10. Lyon, France: International Agency for Research on Cancer; Year 2010 — http://globocan.iarc.fr
- See also: Accessed 08/08/2012 — http://www.seer.cancer.gov
- See also: Ipilimumab or High-Dose Interferon Alfa-2b in Treating Patients With High-Risk Stage III-IV Melanoma That Has Been Removed by Surgery — http://www.clinicaltrials.gov/ct2/show/NCT01274338

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were a total of 39 patients enrolled to this study; 9 participants enrolled to arm A, 16 participants enrolled onto arm B and 14 to C.
Groups:
- Arm B- Nivolumab: Nivolumab administration:
  Three doses of nivolumab will be administered to enrolled patients on Day -42, Day -28, and Day-14 (+/- two days) prior to planned surgery on Day 0 or up to +10 days.
  Nivolumab: Anti-PD-1 Therapy
Period: Overall Study
Arm/Group | Arm A- Nivolumab and Ipilimumab | Arm B- Nivolumab | Arm C- Nivolumab, Carboplatin, & Paclitaxel
Started | 9 | 16 | 14
Completed | 9 | 16 | 14
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A- Nivolumab and Ipilimumab | Arm B- Nivolumab | Arm C- Nivolumab, Carboplatin, & Paclitaxel | Total
Number analyzed (Participants) | 9 | 16 | 14 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 5 | 14
  >=65 years | 5 | 11 | 9 | 25
Age, Continuous [Mean (Full Range); unit: years] | 68 [53 to 84] | 69 [52 to 81] | 68 [46 to 78] | 69 [46 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 8 | 17
  Male | 7 | 9 | 6 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White/Non-Hispanic | 7 | 14 | 10 | 31
  Race/Ethnicity: Black or African American/Unknown | 0 | 1 | 0 | 1
  Race/Ethnicity: White/Declined to answer | 1 | 1 | 0 | 2
  Race/Ethnicity: Unknown/Non-Hispanic | 0 | 0 | 2 | 2
  Race/Ethnicity: American Indian or Alaskan Native/Non-Hispanic | 1 | 0 | 1 | 2
  Race/Ethnicity: Other/Non-Hispanic | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 0 | 2 | 11 | 13
  United States | 9 | 14 | 3 | 26

OUTCOME MEASURES:

1. Primary Outcome: Safety as Measured by Number of Participants With Grade 3 and 4 Lab Abnormalities, as Defined by CTCAE v4.03
Description: Safety will be measured by drawing safety labs. (CBC and a Chemistry Panel will be drawn at 2 week intervals during Nivolumab administration). Grade 3 and 4 lab abnormalities will be recorded from both participating sites.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A- Nivolumab and Ipilimumab | Arm B- Nivolumab | Arm C- Nivolumab, Carboplatin, & Paclitaxel
Number analyzed (Participants) | 9 | 16 | 14
Participants | 1 | 1 | 1

2. Primary Outcome: Safety as Assessed by Number of Grade 3 and 4 Adverse Events
Description: Number of Grade 3 and 4 adverse events as defined by CTCAE v4.03 that occur while a subject is participating in the study.
Time Frame: 8 weeks
Measure: Number; unit: events
Arm/Group | Arm A- Nivolumab and Ipilimumab | Arm B- Nivolumab | Arm C- Nivolumab, Carboplatin, & Paclitaxel
Number analyzed (Participants) | 9 | 16 | 14
events | 1 | 1 | 1

3. Secondary Outcome: Pathologic Response
Description: Pathologic response to neoadjuvant nivolumab, nivolumab plus ipilimumab, and nicvolumab, carboplatin, and paclitaxel in resected tumor and lymph nodes. The rate of major pathologic response, defined as <10% residual viable tumor cells in the resection specimen will be compared to historic data with neoadjuvant chemotherapy.
Time Frame: 6 weeks
Reporting Status: Not Posted, anticipated posting 2026-08

4. Secondary Outcome: Radiographic Response
Description: Radiographic response to neoadjuvant nivolumab, nivolumab plus ipilimumab, and carboplatin and paclitaxel as defined by RECIST 1.1.
Time Frame: 5 weeks
Reporting Status: Not Posted, anticipated posting 2026-08

ADVERSE EVENTS:
Time Frame: From the time of first dose of study medication up to 8 weeks.
Arm/Group | Arm A- Nivolumab and Ipilimumab | Arm B- Nivolumab | Arm C- Nivolumab, Carboplatin, & Paclitaxel
All-Cause Mortality (participants affected / at risk) | 1/9 | 0/16 | 0/14
Serious Adverse Events (participants affected / at risk) | 1/9 | 4/16 | 2/14
Other Adverse Events (participants affected / at risk) | 9/9 | 15/16 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A- Nivolumab and Ipilimumab (N=9) | Arm B- Nivolumab (N=16) | Arm C- Nivolumab, Carboplatin, & Paclitaxel (N=14)
posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
infusion reaction (General disorders) | 0 (0) | 1 (1) | 0 (0)
lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
adult repiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A- Nivolumab and Ipilimumab (N=9) | Arm B- Nivolumab (N=16) | Arm C- Nivolumab, Carboplatin, & Paclitaxel (N=14)
dizziness (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
constipation (Gastrointestinal disorders) | 1 (1) | 4 (4) | 8 (8)
non-cardiac chest pain (General disorders) | 2 (2) | 6 (6) | 0 (0)
neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (6) | 6 (6)
nausea (Gastrointestinal disorders) | 2 (3) | 1 (1) | 6 (6)
anemia (Blood and lymphatic system disorders) | 0 (0) | 4 (4) | 2 (2)
irritability (General disorders) | 0 (0) | 1 (1) | 0 (0)
fatigue (General disorders) | 5 (5) | 6 (6) | 6 (7)
anorexia (Metabolism and nutrition disorders) | 3 (4) | 2 (2) | 7 (8)
lip infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (6) | 1 (1)
wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 3 (4) | 2 (3)
blurred vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
anxiety (Psychiatric disorders) | 3 (3) | 4 (4) | 1 (1)
localized edema (General disorders) | 0 (0) | 1 (1) | 0 (0)
bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
hyperthyroidism (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0)
hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
pruritis (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (2) | 3 (3)
skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | 5 (5)
seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
headache (Nervous system disorders) | 2 (4) | 2 (2) | 1 (1)
dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4) | 1 (1)
peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 4 (4) | 2 (3)
diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3)
blood and lymphatic system disorders - other (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
infusion related reaction (General disorders) | 1 (1) | 1 (1) | 0 (0)
hypertension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
venous injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
depression (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0)
dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (5) | 1 (3)
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0)
insomnia (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0)
hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
mucosal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
paresthesia (Nervous system disorders) | 0 (0) | 1 (1) | 4 (4)
chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 8 (8)
dry cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
arthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (1)
mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 4 (5)
postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
edema limbs (General disorders) | 1 (1) | 0 (0) | 1 (1)
chills (General disorders) | 1 (1) | 0 (0) | 2 (2)
surgical and medical procedures - other (Surgical and medical procedures) | 1 (1) | 0 (0) | 3 (3)
vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
chest pain - cardiac (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
urinary urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
floaters (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
neck edema (General disorders) | 2 (2) | 0 (0) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
recurrent laryngeal nerve palsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-21): https://cdn.clinicaltrials.gov/large-docs/21/NCT02259621/Prot_SAP_003.pdf